CLINICAL TRIAL: NCT00079417
Title: Trial of Systemic Neoadjuvant Chemotherapy for Group B Intraocular Retinoblastoma
Brief Title: Neoadjuvant Carboplatin and Vincristine and Standard Local Ophthalmic Therapy in Treating Patients With Intraocular Retinoblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARET0331; NCI-2009-00422 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARET0331; CDR0000355721; COG-ARET0331; ARET0331 (Other: Children's Oncology Group); ARET0331 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-01

CONDITIONS: Intraocular Retinoblastoma
MeSH Terms: interventions — Carboplatin; Cryosurgery; Iodine-125; Radiotherapy; Radiation; Ruthenium-106; Vincristine

ARMS (1):
- Treatment (chemotherapy, surgery) (Experimental): Patients receive chemoreduction comprising carboplatin IV over 60 minutes followed by vincristine IV over 1-2 minutes on day 1. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. After the first course of chemoreduction, patients undergo standardized local ophthalmic therapy comprising local laser therapy, cryotherapy, and/or radioactive plaque comprising iodine I 125 or ruthenium Ru 106.
  Interventions: Drug: Carboplatin; Procedure: Cryosurgery; Procedure: Infrared Laser Therapy; Radiation: Iodine I-125; Radiation: Radiation Therapy; Radiation: Ruthenium Ru-106; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Cryosurgery
  Other Names: Ablation, Cryo; Cryoablation; cryosurgical ablation
Procedure: Infrared Laser Therapy
Radiation: Iodine I-125 — Undergo radioactive therapy
  Other Names: 125-Iodine; I-125; Iodine 125; Iodine I 125
Radiation: Radiation Therapy — Undergo radioactive therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Radiation: Ruthenium Ru-106 — Undergo radioactive therapy
  Other Names: Ru-106; Ruthenium Ru 106
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase III trial is studying how well giving carboplatin and vincristine together with standard local ophthalmic therapy works in treating children with intraocular retinoblastoma. Drugs used in chemotherapy, such as carboplatin and vincristine, work in different ways to stop tumor from dividing so they stop growing or die. It is not yet known whether neoadjuvant chemotherapy combined with standard local ophthalmic therapy is effective in treating intraocular retinoblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the 2-year event-free survival of patients with Group B intraocular retinoblastoma treated with neoadjuvant chemoreduction comprising carboplatin and vincristine and standardized local ophthalmic therapy.

SECONDARY OBJECTIVES:

I. Determine the response rate after one course of chemoreduction (before standardized local ophthalmic therapy) in these patients.

II. Correlate response rate with event-free survival in patients treated with this regimen.

III. Determine the incidence of toxic effects in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive chemoreduction comprising carboplatin IV over 60 minutes followed by vincristine IV over 1-2 minutes on day 1. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. After the first course of chemoreduction, patients undergo standardized local ophthalmic therapy comprising local laser therapy, cryotherapy, and/or radioactive plaque comprising iodine I 125 or ruthenium Ru 106.

Patients are followed every 3-4 weeks until there is no active tumor seen on a minimum of 3 ophthalmic exams under anesthesia, every 6-8 weeks until 3 years of age, every 4-6 months until 10 years of age, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Group B intraocular retinoblastoma meeting 1 of the following criteria:

  * Group B tumor(s) in 1 eye
  * Group B tumor(s) in both eyes
  * Group A tumor in 1 eye and Group B tumor(s) in the other eye
  * Group E tumor in 1 eye that has been enucleated and Group B tumor(s) in the remaining eye at the time of enucleation of the Group E tumor
* Defined by the International Classification System for Intraocular Retinoblastoma as follows:

  * Group A: Small tumors (≤ 3 mm in greatest dimension) confined to the retina, away from foveola and disc meeting the following criteria:

    * More than 3 mm from fovea
    * More than 1.5 mm from optic disk
  * Group B: Tumors more than 3 mm meeting the following criteria:

    * Confined to the retina in any location not in Group A
    * Tumor associated subretinal fluid < 3 mm from the tumor margin with no subretinal seeding
  * Group E: Must have ≥ 1 of the following present:

    * Tumor touching the lens
    * Tumor anterior to anterior vitreous face involving ciliary body or anterior segment
    * Diffuse infiltrating retinoblastoma
    * Neovascular glaucoma
    * Opaque media from hemorrhage
    * Tumor necrosis with aseptic orbital cellulites
    * Phthisis bulbi
* Confirmation of diagnosis by CT scan or MRI of the brain and orbits AND an ophthalmologic evaluation under anesthesia within the past 3 weeks
* No choroidal and/or optic nerve invasion past the lamina cribosa
* No evidence of extraocular retinoblastoma clinically or by head and orbital MRI and/or CT scan
* No tumor present on histological exam at the cut end of the optic nerve for any Group E eye enucleated before study entry
* Performance status - ECOG 0-2
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* AST or ALT < 2.5 times ULN for age
* Creatinine clearance (based on Schwartz formula) or radioisotope glomerular filtration rate ≥ 70mL/min/1.73 m^2
* No prior chemotherapy
* No other concurrent chemotherapy
* No prior radiotherapy
* No other concurrent radiotherapy, including intensity-modulated stereotactic, or proton beam radiotherapy
* Prior enucleation of one eye allowed provided the remaining eye is Group B
* No concurrent enucleation
* No prior local ophthalmic therapy for retinoblastoma
* No other prior therapy for retinoblastoma
* No local therapy during chemotherapy course 1

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2005-12-26 (Actual); Primary Completion 2010-01-01 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra L Friedman, Principal Investigator — Children's Oncology Group
Locations (10):
- United States (10):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Vincristine Sulfate and Carboplatin and Surgery: Patients receive chemoreduction comprising carboplatin IV (Pts < 36 months: 18.6 mg/kg Pts ≥ 36 months: 560 mg/m2) over 60 minutes followed by vincristine sulfate IV (Pts < 36 months: 0.05 mg/kg Pts ≥36 months: 1.5 mg/m2) over 1-2 minutes on day 1. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. After the first course of chemoreduction, patients undergo standardized local ophthalmic therapy comprising local infrared laser therapy, cryosurgery, and/or radiation therapy (radioactive) plaque comprising iodine I 125 or ruthenium Ru 106.
  cryosurgery: Application of extreme cold to destroy abnormal or diseased tissue.
  infrared laser therapy: Laser therapy or "photobiomodulation" is the use of specific wavelength of light (red and near-infrared) to create therapeutic effects
  iodine I 125: Undergo radioactive therapy
  ruthenium Ru 106: Undergo radioactive therapy
  carboplatin: Given IV
  vincristine sulfate: Given IV
Period: Overall Study
Arm/Group | Vincristine Sulfate and Carboplatin and Surgery
Started | 28
Completed | 19
Not Completed | 9
Not completed — Physician Decision | 2
Not completed — Ineligible | 7

BASELINE CHARACTERISTICS:
Groups:
- Vincristine Sulfate and Carboplatin and Surgery: Patients receive chemoreduction comprising carboplatin IV (Pts < 36 months: 18.6 mg/kg Pts ≥ 36 months: 560 mg/m2) over 60 minutes followed by vincristine sulfate IV (Pts < 36 months: 0.05 mg/kg Pts ≥36 months: 1.5 mg/m2) over 1-2 minutes on day 1. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. After the first course of chemoreduction, patients undergo standardized local ophthalmic therapy comprising local infrared laser therapy, cryosurgery, and/or radiation therapy (radioactive) plaque comprising iodine I 125 or ruthenium Ru 106.
Arm/Group | Vincristine Sulfate and Carboplatin and Surgery
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: Years] | 0.3 [0 to 2.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 19
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 27
  Barbados | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Proportion of patients with event free survival at 2 years. An event is defined as the need for non-protocol therapy, defined as additional on-protocol chemotherapy, enucleation or external beam radiation, among patients with Group B intraocular tumors with a schedule of neoadjuvant 2-agent (Vincristine/Carboplatin) chemotherapy (chemo-reduction) and standardized local ophthalmic therapy.
Time Frame: At 2 years
Population: All eligible patients are reported. 7 patients were excluded due to ineligible status. Of the 7 patients, 1 was determined to have only a Group A involved eye and the other 6 had an intact eye that was Group C or D.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Vincristine Sulfate and Carboplatin and Surgery
Number analyzed (Participants) | 21
Proportion of participants | 0.65 [0.40 to 0.82]

2. Secondary Outcome: Response Rate (RR) at Patient Level After the First Course of Therapy
Description: RR will be estimated. The response after 1 course of chemotherapy will be used to better define response to this neoadjuvant systemic chemotherapy, prior to the use of local ophthalmic therapy. Response to subsequent courses will help define response to combined systemic chemotherapy and local ophthalmic therapy. Number of patients with Type I, II, III or IV response after first course of therapy
Time Frame: 1 month after enrollment
Population: All eligible patients are reported. 7 patients were excluded due to ineligible status.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Vincristine Sulfate and Carboplatin and Surgery
Number analyzed (Participants) | 21
Proportion of participants | 0.71 [0.48 to 0.89]

3. Secondary Outcome: Response Rate (RR) at Eye Levels After the First Course of Therapy
Description: RR will be estimated. The response after 1 course of chemotherapy will be used to better define response to this neoadjuvant systemic chemotherapy, prior to the use of local ophthalmic therapy. Response to subsequent courses will help define response to combined systemic chemotherapy and local ophthalmic therapy. Number eyes with Type I, II, III or IV response after first course of therapy
Time Frame: 1 month after enrollment
Population: Number of Group B eyes for the eligible patients. 4 patients were excluded due to ineligible status.
Measure: Number (95% Confidence Interval); unit: Proportion of eyes
Arm/Group | Vincristine Sulfate and Carboplatin and Surgery
Number analyzed (Participants) | 24
Proportion of eyes | 0.71 [0.49 to 0.87]

4. Secondary Outcome: Event-free Survival Rate (EFSR) Defined as the Need for Non-protocol Chemotherapy, Enucleation, or EBRT at the Patient Level
Description: EFSR will be estimated for patients who respond to vincristine and carboplatin after an initial 1 cycle of chemoreduction
Time Frame: 2 years after enrollment
Population: There were 15 eligible patients who responded to vincristine and carboplatin after an initial 1 cycle of therapy. 7 patients were excluded due to ineligible status.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Vincristine Sulfate and Carboplatin and Surgery
Number analyzed (Participants) | 15
Proportion of participants | 0.60 [0.40 to 0.91]

5. Secondary Outcome: Toxicity as Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0
Description: Participants with Grade 3 and higher reported on protocol therapy
Time Frame: 6 months after enrollment
Population: All eligible patients are reported. 7 patients were excluded due to ineligible status.
Measure: Number; unit: Participants
Arm/Group | Vincristine Sulfate and Carboplatin and Surgery
Number analyzed (Participants) | 21
Participants
  Incidence of Catheter Related Infection | 1
  Incidence of Upper Respiratory Infection | 1
  Incidence of Dehydration | 1
  Incidence of Urticaria | 1
  Incidence of Neutrophils | 6

ADVERSE EVENTS:
Description: Adverse events grade 3 and above were considered as Serious Adverse Events in this study. All eligible patients are reported.
Arm/Group | Vincristine Sulfate and Carboplatin and Surgery
Serious Adverse Events (participants affected / at risk) | 10/21
Other Adverse Events (participants affected / at risk) | 3/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vincristine Sulfate and Carboplatin and Surgery (N=21)
Catheter related infection (Infections and infestations) | 1 — Grades 3-5
Dehydration (Metabolism and nutrition disorders) | 1 — Grades 3-5
Neutrophil count decreased (Investigations) | 6 — Grades 3-5
Upper respiratory infection (Infections and infestations) | 1 — Grades 3-5
Urticaria (Skin and subcutaneous tissue disorders) | 1 — Grades 3-5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vincristine Sulfate and Carboplatin and Surgery (N=21)
Neutrophil count decreased (Investigations) | 1 — Grades 1-2
Platelet count decreased (Investigations) | 2 — Grades 1-2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.